CLINICAL TRIAL: NCT02565108
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study to Investigate Possible Drug-drug Interactions Between Clobazam and Cannabidiol (GWP42003-P)
Brief Title: A Randomized Controlled Trial to Investigate Possible Drug-drug Interactions Between Clobazam and Cannabidiol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1428 Blinded Phase; 2014-002942-33 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
Keywords: Cannabidiol; GWP42003-P; Clobazam; Epidiolex; CBD
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol; Clobazam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GWP42003-P 20 mg/kg/Day Dose (Experimental): Participants received GWP42003-P 20 milligrams [mg]/kilogram [kg]/day orally, twice daily immediately after their clobazam (CLB) dose. Participants titrated GWP42003-P to 20 mg/kg/day over 10 days and remained at this dose for the 21-day treatment period. Participants who then did not enter the open-label extension (OLE) or withdrew early had a 10-day taper (10% per day) period. Participants who transferred to the OLE (still blinded at that stage) tapered off their GWP42003-P treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P for the OLE.
  All participants (in the GWP42003-P and Placebo treatment groups) were on a stable dose of CLB at Baseline, administered either once or twice daily as per the physician's preferred CLB dosing regimen for each participant, and continued taking CLB, as an Investigational Medicinal Product (IMP), for the duration of this study.
  Interventions: Drug: GWP42003-P 20 mg/kg/Day Dose; Drug: Clobazam
- Placebo (Placebo Comparator): Participants received placebo (0 mg/milliliter [mL] GWP42003-P) orally, twice daily immediately after the participant's CLB dose. Participants titrated the placebo dose over 10 days, followed by a 21-day treatment period. Participants who then did not enter the OLE or withdrew early had a 10-day taper (10% per day) period. Participants who transferred to the OLE (still blinded at that stage) tapered off their placebo treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P for the OLE.
  All participants (in the GWP42003-P and Placebo treatment groups) were on a stable dose of CLB at Baseline, administered either once or twice daily as per the physician's preferred CLB dosing regimen for each participant, and continued taking CLB, as an IMP, for the duration of this study.
  Interventions: Drug: Placebo; Drug: Clobazam

INTERVENTIONS:
Drug: GWP42003-P 20 mg/kg/Day Dose — GWP42003-P was an oral solution containing 25 mg/mL cannabidiol (CBD) or 100 mg/mL CBD dissolved in the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Other Names: CBD; Cannabidiol; Epidiolex
  Arms: GWP42003-P 20 mg/kg/Day Dose
Drug: Placebo — Placebo oral solution contained the excipients sesame oil and anhydrous ethanol (79 mg/mL) with added sweetener (0.5 mg/mL sucralose) and strawberry flavoring (0.2 mg/mL).
  Arms: Placebo
Drug: Clobazam — Participants were already on a stable dose of CLB at Baseline and continued to take a stable dose of CLB for the duration of the blinded phase of the study. CLB was administered either once or twice daily in line with the physician's preferred dosing regimen for the CLB for each participant.
  Other Names: CLB

SUMMARY:
This trial consists of 2 parts: a double-blinded phase and an open-label extension phase. The blinded phase only will be described in this record. Participants were randomized in a 4:1 ratio to receive GWP42003-P or matching placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have had epilepsy, as determined by the investigator, and must have been taking CLB.
* Participant must have had a documented magnetic resonance imaging/computerized tomography of the brain ruling out a progressive neurologic condition.
* Participant must have experienced at least 1 seizure of any type (that is, convulsive: tonic-clonic, tonic, clonic, atonic; focal: focal seizures with retained consciousness and a motor component, focal seizures with impaired consciousness, focal seizures evolving to bilateral secondary generalization) within the 2 months prior to randomization.
* Participant must have been taking CLB and no more than 2 other antiepileptic drugs (AEDs) during the course of the trial.
* AED(s), including CLB, must have been stable for 4 weeks prior to screening and regimen must have remained stable throughout the duration of the blinded phase of the trail.
* Intervention with vagus nerve stimulation and/or ketogenic diet must be stable for 4 weeks prior to Baseline and participant/caregiver must have been willing to maintain a stable regimen throughout the blinded phase of the study.

Key Exclusion Criteria:

* Participant had clinically significant unstable medical conditions other than epilepsy.
* Participants were on CLB at doses above 20 mg per day.
* Participants taking CLB intermittently as rescue medication.
* Participant had a history of symptoms related to a drop in blood pressure due to postural changes (for example, dizziness, light-headedness, blurred vision, palpitations, weakness, syncope).
* Participant had any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale in the last month or at screening.
* Participant had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to screening or enrollment, other than epilepsy.
* Participant had consumed alcohol during the 7 days prior to enrollment and was unwilling to abstain during the blinded phase of the trail.
* Participant was currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to trial entry.
* Participant had any known or suspected history of any drug abuse or addiction.
* Participant was unwilling to abstain from recreational or medicinal cannabis, or synthetic cannabinoid based medications (including Sativex) for the duration for the study.
* Participant consumed grapefruit or grapefruit juice 7 days prior to enrollment and was unwilling to abstain from drinking grapefruit juice within 7 days of pharmacokinetic visits.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP, for example, sesame oil.
* Participant received an IMP within the 12 weeks prior to the screening visit.
* Participant had significantly impaired hepatic function at the screening or randomization visit, defined as any of the following:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN).
  * ALT or AST > 3 × ULN and total bilirubin > 2 × ULN or international normalized ratio > 1.5.
  * ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Barcelona, Spain
- United Kingdom (4):
  - Birmingham
  - Brighton
  - Leeds
  - Salford

REFERENCES:
- [Derived] VanLandingham KE, Crockett J, Taylor L, Morrison G. A Phase 2, Double-Blind, Placebo-Controlled Trial to Investigate Potential Drug-Drug Interactions Between Cannabidiol and Clobazam. J Clin Pharmacol. 2020 Oct;60(10):1304-1313. doi: 10.1002/jcph.1634. Epub 2020 Jul 11. PMID 32652616

RESULTS

PARTICIPANT FLOW:
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received GWP42003-P 20 milligrams (mg)/kilogram (kg)/day orally, twice daily immediately after their clobazam (CLB) dose. Participants titrated GWP42003-P to 20 mg/kg/day over 10 days and remained at this dose for the 21-day treatment period. Participants who then did not enter the open-label extension (OLE) or withdrew early had a 10-day taper (10% per day) period. Participants who transferred to the OLE (still blinded at that stage) tapered off their GWP42003-P treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P for the OLE.
  All participants (in the GWP42003-P and Placebo treatment groups) were on a stable dose of CLB at Baseline, administered either once or twice daily as per the physician's preferred CLB dosing regimen for each participant, and continued taking CLB, as an Investigational Medicinal Product (IMP), for the duration of this study.
Period: Overall Study
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Started (Randomized) | 16 | 4
Safety Set (Received at least 1 IMP dose; analyzed as treatment received.) | 16 | 4
Pharmacokinetic (PK) Set (Received at least 1 IMP dose, had not reduced CLB dose between Days 1 and 33, and provided PK data.) | 10 | 3
Completed | 14 | 4
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received a dose of GWP42003-P or placebo.
Groups:
- GWP42003-P 20 mg/kg/Day Dose: Participants received GWP42003-P 20 mg/kg/day orally, twice daily immediately after their CLB dose. Participants titrated GWP42003-P to 20 mg/kg/day over 10 days and remained at this dose for the 21-day treatment period. Participants who then did not enter the OLE or withdrew early had a 10-day taper (10% per day) period. Participants who transferred to the OLE (still blinded at that stage) tapered off their GWP42003-P treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P for the OLE.
  All participants (in the GWP42003-P and Placebo treatment groups) were on a stable dose of CLB at Baseline, administered either once or twice daily as per the physician's preferred CLB dosing regimen for each participant, and continued taking CLB, as an IMP, for the duration of this study.
- Placebo: Participants received placebo (0 mg/mL GWP42003-P) orally, twice daily immediately after the participant's CLB dose. Participants titrated the placebo dose over 10 days, followed by a 21-day treatment period. Participants who then did not enter the OLE or withdrew early had a 10-day taper (10% per day) period. Participants who transferred to the OLE (still blinded at that stage) tapered off their placebo treatment by reducing their maintenance dose by 10% per day and concomitantly titrating GWP42003-P for the OLE.
  All participants (in the GWP42003-P and Placebo treatment groups) were on a stable dose of CLB at Baseline, administered either once or twice daily as per the physician's preferred CLB dosing regimen for each participant, and continued taking CLB, as an IMP, for the duration of this study.
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo | Total
Number analyzed (Participants) | 16 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.60 (8.51) | 37.57 (10.67) | 36.79 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Measured Plasma Concentration (Cmax) Of CLB And N-CLB With GWP42003-P Treatment, Days 1 And 33
Description: The Cmax of CLB and its primary metabolite N-desmethylclobazam (N-CLB) was measured on Day 1 (before beginning GWP42003-P treatment; participants were taking CLB only) and Day 33 (following 21 days of GWP42003-P or placebo maintenance; participants were taking CLB and GWP42003-P or CLB and placebo). PK samples were taken at time points relative to the morning dose of CLB, as follows: Predose, 15 minutes (min), 30 min, 1 hour (h), 1.5 h, 2 h, 4 h, 6 h, 12 h, and 24 h.
  One participant in the placebo group was excluded from the PK set because placebo was administered on Day 1, after predose sampling. Six participants in the GWP42003-P group were excluded from the PK set because of GWP42003-P and/or CLB dose modification, discontinuation of IMP, discontinuation from trial, or administration of incorrect IMP dose.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 h postdose on Days 1 and 33
Population: PK Set: All participants who received at least 1 dose of GWP42003-P or placebo, who had not reduced their CLB dose between Day 1 and Day 33, and who provided some on-treatment data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 3
ng/mL
  Cmax: CLB Day 1 | 330 (40.4) | 440 (29.9)
  Cmax: CLB Day 33 | 329 (54.8) | 461 (102.3)
  Cmax: N-CLB Day 1 | 2060 (138.4) | 1130 (82.1)
  Cmax: N-CLB Day 33 | 4570 (54.0) | 1320 (134.1)
  Cmax: CLB Dose-normalized Day 1 | 19.3 (31.4) | 22.0 (29.9)
  Cmax: CLB Dose-normalized Day 33 | 19.2 (44.7) | 23.1 (102.3)
  Cmax: N-CLB Dose-normalized Day 1 | 121 (125.1) | 56.6 (82.1)
  Cmax: N-CLB Dose-normalized Day 33 | 267 (38.6) | 66.1 (134.1)

2. Primary Outcome: PK: Time To The Maximum Plasma Concentration (Tmax) Of CLB And N-CLB With GWP42003-P Treatment, Days 1 And 33
Description: The tmax of CLB and its primary metabolite N-CLB was measured on Day 1 (before beginning GWP42003-P treatment; participants were taking CLB only) and Day 33 (following 21 days of GWP42003-P or placebo maintenance; participants were taking CLB and GWP42003-P or CLB and placebo). PK samples were taken at time points relative to the morning dose of CLB, as follows: Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 12 h, and 24 h.
  One participant in the placebo group was excluded from the PK set because placebo was administered on Day 1, after predose sampling. Six participants in the GWP42003-P group were excluded from the PK set because of GWP42003-P and/or CLB dose modification, discontinuation of IMP, discontinuation from trial, or administration of incorrect IMP dose.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 h postdose on Days 1 and 33
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 3
h
  tmax: CLB Day 1 | 1.00 [0.8 to 4.0] | 1.17 [1.0 to 1.5]
  tmax: CLB Day 33 | 1.86 [0.5 to 4.0] | 1.58 [1.5 to 2.0]
  tmax: N-CLB Day 1 | 1.50 [0.3 to 6.0] | 2.00 [0.0 to 12.0]
  tmax: N-CLB Day 33 | 3.03 [0.0 to 11.1] | 1.00 [0.3 to 2.0]

3. Primary Outcome: PK: Area Under The Plasma Concentration-Time Curve Over A Dosing Interval, Where Tau Is The Dosing Interval (AUCtau) Of CLB And N-CLB With GWP42003-P Treatment, Days 1 And 33
Description: The AUCtau of CLB and its primary metabolite N-CLB was measured on Day 1 (before first GWP42003-P dose; participants were taking CLB only) and Day 33 (following 21 days of GWP42003-P or placebo maintenance; participants were taking CLB and GWP42003-P or CLB and placebo). PK samples were taken at time points relative to the morning dose of CLB, as follows: Predose, 15 min, 30 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, 12 h, and 24 h.
  One participant in the placebo group was excluded from the PK set because placebo was administered on Day 1, after predose sampling. Six participants in the GWP42003-P group were excluded from the PK set because of GWP42003-P and/or CLB dose modification, discontinuation of IMP, discontinuation from trial, or administration of incorrect IMP dose.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 h postdose on Days 1 and 33
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 3
h*ng/mL
  AUCtau: CLB Day 1 | 2690 (52.9) | 3320 (67.5)
  AUCtau: CLB Day 33 | 2840 (46.2) | 3310 (102.5)
  AUCtau: N-CLB Day 1 | 18300 (124.2) | 11400 (63.7)
  AUCtau: N-CLB Day 33 | 48400 (53.9) | 11500 (79.1)
  AUCtau: CLB Dose-normalized Day 1 | 157 (47.1) | 166 (67.5)
  AUCtau: CLB Dose-normalized Day 33 | 166 (34.7) | 165 (102.5)
  AUCtau: N-CLB Dose-normalized Day 1 | 1070 (105.1) | 571 (63.7)
  AUCtau: N-CLB Dose-normalized Day 33 | 2830 (38.3) | 573 (79.1)

4. Primary Outcome: PK: Geometric Mean Ratios Of CLB And N-CLB For Cmax On Day 33 Compared With Day 1
Description: The Day 33 compared to Day 1 geometric mean ratios of CLB and N-CLB were calculated for Cmax to look for evidence of drug-drug interactions between GWP42003-P/Placebo and CLB and between GWP42003-P/Placebo and N-CLB. A standard 90% confidence interval (CI) approach for the between time point ratios of geometric means of Cmax was carried out on a logarithmic scale using a linear mixed effect model. The no-effect boundary was set between 0.5 and 2.0, and if the 90% CI for the ratio of the geometric means of a PK variable fell within the interval [0.5, 2.0], a lack of meaningful effect was declared. Estimates were back transformed to provide summaries on the original scale. The model included a fixed effect term for PK assessment period. An unstructured covariance matrix was used. Kenward and Roger's method was used to calculate the denominator degrees of freedom for the fixed effects.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 h postdose on Days 1 and 33
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 3
Ratio
  Geometric Mean Ratio of CLB, Cmax | 0.997 [0.834 to 1.19] | 1.05 [0.401 to 2.74]
  Geometric Mean Ratio of N-CLB, Cmax | 2.22 [1.42 to 3.46] | 1.17 [0.628 to 2.17]

5. Secondary Outcome: Number Of Participants Who Experienced Severe Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event with an onset date on or after the first dose of IMP. If an adverse event (AE) had a partial onset date and it was unclear from the partial date (or the stop date) whether the AE started prior to or following the first dose of IMP then the AE was considered a TEAE. The number of participants who experienced 1 or more severe TEAEs after screening up to Day 71.
  A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Postdose on Day 2 up to Safety follow-up (Day 71)
Population: Safety Set: all participants who received at least 1 dose of IMP (GWP42003-P or placebo). Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 16 | 4
Participants | 1 | 0

6. Primary Outcome: PK: Geometric Mean Ratios Of CLB And N-CLB For AUCtau On Day 33 Compared With Day 1
Description: The Day 33 compared to Day 1 geometric mean ratios of CLB and N-CLB were calculated for AUCtau to look for evidence of drug-drug interactions between GWP42003-P/Placebo and CLB and between GWP42003-P/Placebo and N-CLB. A standard 90% CI approach for the between time point ratios of geometric means of AUCtau was carried out on a logarithmic scale using a linear mixed effect model. The no-effect boundary was set between 0.5 and 2.0, and if the 90% CI for the ratio of the geometric means of a PK variable fell within the interval [0.5, 2.0], a lack of meaningful effect was declared. Estimates were back transformed to provide summaries on the original scale. The model included a fixed effect term for PK assessment period. An unstructured covariance matrix was used. Kenward and Roger's method was used to calculate the denominator degrees of freedom for the fixed effects.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 12, and 24 h postdose on Days 1 and 33
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Number analyzed (Participants) | 10 | 3
Ratio
  Geometric Mean Ratio of CLB, AUCtau | 1.06 [0.898 to 1.24] | 0.996 [0.652 to 1.52]
  Geometric Mean Ratio of N-CLB, AUCtau | 2.64 [1.95 to 3.58] | 1.00 [0.795 to 1.27]

ADVERSE EVENTS:
Time Frame: Following screening up to Day 71
Description: The safety analysis set included all participants randomized to treatment who received at least 1 dose of IMP. Participant data were analyzed according to the treatment they received.
Arm/Group | GWP42003-P 20 mg/kg/Day Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/4
Other Adverse Events (participants affected / at risk) | 12/16 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=16) | Placebo (N=4)
Seizure cluster (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GWP42003-P 20 mg/kg/Day Dose (N=16) | Placebo (N=4)
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Sedation (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0
Tearfulness (Psychiatric disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1/8 | 0/2
Seasonal allergy (Immune system disorders) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days